CLINICAL TRIAL: NCT03212417
Title: Pilot/Feasibility Study of a Compassion Fatigue Education Intervention in Hematology/Oncology Clinical Research Nurses (CRNs) and Bone Morrow Transplant (BMT) Nurses
Brief Title: Education as an Intervention of Compassion Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 17181
Record Dates: First submitted 2017-06-29; First posted 2017-07-11 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Normal Volunteer
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional trial without phases-supportive care. (Other): This is a feasibility pilot study project assessing the presence of compassion fatigue in clinical research nurses (cohort 1) and bone marrow transplant nurses (cohort 2). A survey will be completed by participants prior to and after an educational presentation. The intervention includes the risk factors, signs and symptoms, and interventions on compassion fatigue. The survey will be completed prior to the education, immediately following the education, one month following the education and two months following the education. A final survey will be implemented for the cohort 2 only. The objective of this concluding analysis is to gather data relative to CF and coping mechanisms.
  Interventions: Other: Educational intervention

INTERVENTIONS:
Other: Educational intervention — Presentation of risk factors, signs and symptoms, and interventions on compassion fatigue

SUMMARY:
The purpose of this study is to evaluate the impact education has on reducing compassion fatigue in Oncology Clinical Research Nurses.

DETAILED DESCRIPTION:
Slatten, Carson, and Carson (2011) describe compassion fatigue as "an occupational hazard for those in the helping professions and is a natural consequence of working with people who have experienced extremely stressful events" (p. 327). Compassion fatigue (CF) is a condition that can affect one's physical, emotional, and social well-being. CF can exist or be misunderstood as burnout, defined as the "inability to cope with job stress, displays symptoms such as emotional exhaustion, and reduced personal and professional accomplishments" (Maslach, Schaufeli, & Leiter, 2001). The term Secondary Traumatic stress has been used within the literature to describe nurses' exposure to the traumatic situations of patients and is often used interchangeably with compassion fatigue (Beck, 2011; Flarity, Gentry, & Mesinkoof, 2013), but is contrasted by compassion satisfaction (CS): the pleasure that nurses derive from the ability to perform work well (Stamm, 2009). Slatten et al., (2011) described compassion fatigue as a natural consequence of nursing: therefore, prevention of exposure should not be the focus of any intervention. The Literature review has identified that nurses should be educated about risk factors and coping strategies to combat compassion fatigue.

Neville and Cole (2013) describe incentives for organizations to proactively prevent CF, they explained:

The care patients receive from nurses is one of the most significant predictors of patient satisfaction and is a quality indicator of overall healthcare performance. Research demonstrates that nurses' perception of work environment and patient satisfaction are highly correlated; thus, measures to enhance nurses' ability to deliver excellent care and to thrive in their work environments are of paramount importance to healthcare institutions (p. 349).

Most patients on clinical trials have tried standard of care treatment unsuccessfully. Little is known, due to the lack of research, demonstrating the impact of CF, CS or Burnout on CRNs and BMT Nurses. Both nursing populations' work closely with oncology patients, either during or following participation on a clinical trial, developing a close relationship with the patients and their families. The nurses are at risk for exposure to emotionally disturbing patient outcomes that can be detrimental on psychological health. One-third of the Hematology and Solid Tumor clinical trials at City of Hope National Medical Center are phase 1 trials, which are to determine dose limiting toxicity with the intent of improving patient outcomes. Nurses are providing patient care to individuals with a poor prognosis, after repeat exposure to emotional pain, the CRN and BMT Nurse leave the organization due to intolerance of suffering.

This project is important to teach nurses how to recognize and manage CF. The educational intervention could reduce nurse turnover, increase morale, and improve patient satisfaction, all of which could be a cost savings to the organization.

ELIGIBILITY:
Inclusion Criteria:

* Documented written informed consent of participant
* Must be a Clinical Research Nurse working in the Clinical Trials Office or a Bone Marrow Transplant nurse working at COH National Medical Center
* Ability read and speak English, (questionnaires are in English)
* Willingness and ability to complete three ProQol 5 surveys, one demographic survey,and Coping Mechanisms survey (cohort 2).
* Willingness to participate in a 30-minute educational intervention.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Participation in intervention (Yes/No) | Two months post intervention
Participation in intervention and ProQoL survey (Professional Quality of Life: Compassion and Satisfaction Fatigue Version 5) at one-month and two-month assessment (Yes/No) Coping Mechanisms survey. | Three months post intervention

SECONDARY OUTCOMES:
Descriptive analysis on participant's data collected by demographic information form, including | Three months post intervention
  * Age (categorical, number of participants and percentage):
  * Gender (categorical, number of participants and percentage):
  * Years of RN (categorical, number of participants and percentage):
  * Years of Clinical Research Nurse or Bone Marrow Transplant nurse (categorical, number of participants and percentage):
  * Years of RN at COH (categorical, number of participants and percentage):
  * Years of oncology RN (categorical, number of participants and percentage):
  * Highest level of nursing education (categorical, number of participants and percentage)
  * Ethnicity (categorical, number of participants and percentage)
  * Religious preference (categorical, number of participants and percentage)
  * Annual household income (categorical, number of participants and percentage)
  * Marital status (categorical, number of participants and percentage)
Descriptive analysis (median and range) on participant's ProQol score collected by ProQol survey (Professional Quality of Life: Compassion and Satisfaction Fatigue Version 5) at the intervention, one-month, and two-month assessment. | From intervention to two-month post intervention
Calculate the changes of ProQol score from intervention to one-month post intervention | From intervention to one-month post intervention
Calculate the changes of ProQol score from intervention to two-month post intervention | From intervention to two-month post intervention
Descriptive analysis (median and range) on participant's coping mechanisms score collected at the three-month post intervention | From intervention to three-month post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lynette Svingen, MBA/MHA, RN, BSN, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No